CLINICAL TRIAL: NCT04649333
Title: COVID-19 and Sports - an Online Survey on the Impact of the Pandemic and Possible Preventive Measures
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Collaborators: Universitaet Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 20200609
Record Dates: First submitted 2020-11-30; First posted 2020-12-02 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study was to investigate the effects of the COVID-19 pandemic on individual and general sport activities in an effort to provide information for safe return to community sports.

ELIGIBILITY:
Inclusion Criteria:

-Age over 18 years

Exclusion Criteria:

* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The survey was shared and promoted by the participating universities, some sport organisations and administrators, and by multiple medical colleagues and athletes.
Sampling Method: Non-Probability Sample
Enrollment: 1336 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The type, extent and intensity of physical activity | 10 to15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided